CLINICAL TRIAL: NCT05832151
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy and Safety of CIN-102 (Deudomperidone) in Adult Subjects With Diabetic Gastroparesis
Brief Title: A Study to Evaluate the Efficacy and Safety of CIN-102 (Deudomperidone) in Adults With Diabetic Gastroparesis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CinDome Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIN-102-123
Record Dates: First submitted 2023-03-16; First posted 2023-04-27 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-08

CONDITIONS: Diabetic Gastroparesis
Keywords: Gastroparesis; Diabetic gastroparesis; Gastrointestinal disease; Delayed gastric emptying; Digestive system diseases; Nausea; Vomiting; Stomach; Dopamine receptor antagonist
MeSH Terms: conditions — Gastroparesis; Gastrointestinal Diseases; Digestive System Diseases; Nausea; Vomiting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CIN-102: Dose 15mg or 10mg (Experimental): CIN-102, Dose 15 mg or 10 mg, twice daily for 12 weeks
  Interventions: Drug: CIN-102 Dose 15mg or 10mg
- Placebo (Placebo Comparator): Placebo for CIN-102, twice daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CIN-102 Dose 15mg or 10mg — 2 capsules twice daily for 12 weeks
  Arms: CIN-102: Dose 15mg or 10mg
Drug: Placebo — 2 capsules twice daily for 12 weeks
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate if the study drug CIN-102 (deudomperidone) can help reduce the symptoms associated with diabetic gastroparesis in adult patients.

The main questions it aims to answer are:

* To evaluate the efficacy of CIN-102 on symptoms of gastroparesis when given to patients with diabetic gastroparesis compared to a placebo
* To evaluate the safety and tolerability of CIN-102 when given to patients with diabetic gastroparesis compared to a placebo

Participants will go through the following schedule:

* Screening period (1-2 visits)
* Lead-in period (1 visit)

  * Will complete a Gastric Emptying Breath Test (GEBT)
  * Will complete daily diary and other Patient Reported Outcomes (PROs) as described in the protocol to assess eligibility for continued study participation
* 12-week treatment period (7 visits)

  * Study drug taken twice daily by mouth
  * Will complete daily diaries and other PROs as described in protocol
* 1 week follow-up (1 visit)

Researchers will compare the effects of the following treatments:

* Drug- CIN-102 Dose 15 mg or 10 mg
* Drug- Placebo

ELIGIBILITY:
Key Inclusion Criteria:

* Is a male or female ≥18 years of age;
* Has a diagnosis of Type 1 or Type 2 diabetes, according to the American Diabetes Association criteria;
* Has a current diagnosis of diabetic gastroparesis defined by the following:

  1. Persistent gastrointestinal symptoms that in the opinion of the Investigator are consistent with gastroparesis within 6 months prior to Screening; AND
  2. Documented delayed gastric emptying as determined by gastric emptying breath test (GEBT), scintigraphy, or manometry.
* Body mass index (BMI) between 18 and 49 kg/m2, inclusive;
* Glycosylated hemoglobin (HbA1c) level <10% at Screening;
* If receiving treatment with GLP-1RA, may be considered for the study if all of the following criteria are satisfied:

  1. The GLP-1 RA has been prescribed for the management of diabetes and not specifically for weight loss/weight management;
  2. Has been on a stable dose of GLP-1RA for a minimum of 3 months before Screening and is anticipated to sustain the same dose during GEBT and throughout the study;
  3. Is tolerating the GLP-1RA well based on Investigator's judgment;
  4. None of the study-qualifying signs/symptoms of gastroparesis are solely attributable to the use of GLP-1RA; and
  5. The symptoms of gastroparesis preceded the initiation of GLP-1RA therapy.
* Willing to washout from ongoing treatment for gastroparesis.

Key Exclusion Criteria:

* Has known cause of gastroparesis other than diabetes (eg, idiopathic gastroparesis and/or gastroparesis attributed to surgery, viral illness, cancer, scleroderma, or other neurologic disorder);
* Has been hospitalized within 3 months prior to Visit 1 for diabetic gastroparesis and/or diabetic ketoacidosis and/or malnutrition;
* History or evidence of clinically significant arrhythmia;
* History of pyloroplasty, pyloromyotomy, or gastric peroral endoscopic myotomy, fundoplication, gastrectomy, vagotomy, or bariatric surgery;
* Currently receiving parenteral feeding or presence of a nasogastric or other enteral tube for feeding or decompression;
* Pyloric injection of botulinum toxin within 6 months of Screening;
* Positive test for drugs of abuse;
* Has a known allergy to eggs or spirulina;
* Females who are pregnant, breastfeeding, or planning to become pregnant or breastfeed during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2025-11-14 (Actual); Study Completion 2025-12-12 (Actual)

PRIMARY OUTCOMES:
Effect of CIN-102 to significantly decrease gastroparesis-related symptoms as compared to baseline based on the composite of the average ANMS GCSI-DD Nausea Sub-Scale and Vomiting Scores | Over the last 2 weeks of the 12-week Treatment Period as compared to baseline
  The American Neurogastroenterology and Motility Society Gastroparesis Cardinal Symptom Index Daily Diary (ANMS GCSI-DD) Nausea Subscale scores and the Vomiting subscale scores will be averaged into a single value that ranges 0-4 (0 for no symptom and 4 for very severe)

SECONDARY OUTCOMES:
Incidence of clinically significant changes, in the Investigator's opinion, in laboratory parameters, physical examination findings, 12-lead ECG parameters, weight measurement. | Over the 12-week Treatment Period
Incidence of treatment-emergent adverse events (TEAEs) | Over the 12-week Treatment Period
Incidence of treatment emergent Serious Adverse Events (SAEs) | Over the 12-week Treatment Period
Incidence of TEAEs leading to premature discontinuation of study drug | Over the 12-week Treatment Period
Incidence of treatment-emergent marked laboratory abnormalities. | Over the 12-week Treatment Period
Percentage of responders who demonstrate an average ≥0.5 reduction from baseline on the ANMS GCSI-DD Nausea Sub-Scale and Vomiting Scores | Over the last 2 weeks of the 12-week Treatment Period
Percentage of subjects achieving a ≥30% reduction from baseline on a composite of the average ANMS GCSI-DD Nausea Sub-Scale and Vomiting Scores | Over the last 2 weeks of the 12-week Treatment Period
The percentage of symptom-free days in the ANMS GCSI-DD Total Score, a composite of the Nausea Sub-Scale and Vomiting Scores, and Sub-Scale Scores | Over the last 2 weeks of the 12-week Treatment Period
  Symptomatic days defined as >mild (ANMS GCSI-DD scores >2)
The relationship between ANMS GCSI-DD Nausea Sub-Scale and Vomiting Scores and Patient Global Impression of Severity (PGIS) and Patient Global Impression of Change (PGIC) over the 12-week Treatment Period; | Over the 12-week Treatment Period
Percentage of subjects with a history of a lack of response or who could not tolerate metoclopramide therapy or other prokinetics, who demonstrate a >30% reduction from baseline on a composite score | Over the last 2 weeks of the 12-week Treatment Period as compared to baseline
  Composite of the average ANMS GCSI-DD Nausea Sub-Scale and Vomiting Scores
Effect of CIN-102 to significantly decrease the severity of gastroparesis-related symptoms as compared to baseline | Over the last 2 weeks of the 12-week Treatment Period as compared to baseline
  Based on the average ANMS GCSI-DD Total and Sub-Scale Scores
The change in the composite of the average ANMS GCSI-DD Nausea Sub-Scale and Vomiting Scores among subjects receiving glucagon-like peptide-1 receptor agonist (GLP-1RA) | Over the 12-week Treatment Period as compared to baseline
The percentage of responders among subjects receiving GLP-1RA who demonstrate an average ≥0.5 reduction from baseline on the ANMS GCSI-DD Nausea Sub-Scale and Vomiting Scores | Over the last 2 weeks of the 12-week Treatment Period
The percentage of subjects receiving GLP-1RA who achieve a ≥30% reduction from baseline on the ANMS GCSI-DD Nausea Sub-Scale and Vomiting Scores | Over the last 2 weeks of the 12-week Treatment Period
The change in the ANMS GSCI-DD Total Score and a composite of gastroparesis-related symptoms among subjects receiving GLP-1RA; | over the last 2 weeks of the 12-week Treatment Period, as compared to baseline
All endpoints that are evaluated over the last 2 weeks of the 12-week Treatment period will also be evaluated over the last 6 weeks of the 12-week Treatment period. | Over the last 6 weeks of the 12-week Treatment Period
Change in the PGIS with each dose of CIN-102 | From baseline to Week 12
Change in the PGIC with each dose of CIN-102 | From baseline to Week 12

CONTACTS AND LOCATIONS:
Locations (100):
- United States (100):
  - Digestive Health Specialists of the Southeast, Dothan, Alabama
  - G & L Research, LLC, Foley, Alabama
  - Clinical Research Associates, LLC, Huntsville, Alabama
  - Phoenix Medical Research Institute, LLC, Peoria, Arizona
  - Onyx Clinical Research, Phoenix, Arizona
  - Del Sol Research Management, LLC, Tucson, Arizona
  - Preferred Research Partners, Inc., Little Rock, Arkansas
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - Arkansas Gastroenterology - North Little Rock, North Little Rock, Arkansas
  - Alliance Research Institute - Bell Gardens, Bell Gardens, California
  - Hope Clinical Research LLC, Canoga Park, California
  - Alliance Research Institute, LLC, Canoga Park, California
  - Erick H. Alayo Medical Corporation, Chula Vista, California
  - GW Research Inc., Chula Vista, California
  - Kindred Medical Institute for Clinical Trials, LLC, Corona, California
  - New Hope Research Development, Corona, California
  - Aurora Care Clinic, Costa Mesa, California
  - Paragon Rx Clinical, Garden Grove, California
  - Valley View Wellness and Medical Center - VVCRD, Garden Grove, California
  - Torrance Clinical Research Institute Inc., Lomita, California
  - Angel City Research, Los Angeles, California
  - Facey Medical Research, Mission Hills, California
  - Millennium Clinical Trials, Thousand Oaks, California
  - Innovative Research of West Florida, Clearwater, Florida
  - USA and International Research Inc., Doral, Florida
  - Advanced Medical Research Group, Hollywood, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - ClinCloud LLC, Maitland, Florida
  - A+ Research Inc, Miami, Florida
  - International Research Associates LLC - Breton, Miami, Florida
  - Advanced Research Institute Inc, New Port Richey, Florida
  - Gastroenterology of Greater Orlando, Orange City, Florida
  - Tandem Clinical Research - Viera, Viera, Florida
  - Summit Clinical Research, LLC, Athens, Georgia
  - Atlanta Center for Gastroenterology P.C., Decatur, Georgia
  - Medisphere Medical Research Center, Evansville, Indiana
  - Lutheran Medical Group, Fort Wayne, Indiana
  - University of Kansas Medical Center (KUMC), Kansas City, Kansas
  - DelRicht Clinical Research - Overland Park, Overland Park, Kansas
  - Kansas Medical Clinic, P.A., Topeka, Kansas
  - Alliance for Multispecialty Research - Wichita West, Wichita, Kansas
  - University of Louisville, Louisville, Kentucky
  - DelRicht Clinical Research - Louisville, Louisville, Kentucky
  - Delta Research Partners, Bastrop, Louisiana
  - Tandem Clinical Research GI - Houma, Houma, Louisiana
  - Tandem Clinical Research, Marrero, Louisiana
  - Tandem Clinical Research GI - Metairie, Metairie, Louisiana
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Aa Mrc, Llc, Flint, Michigan
  - Clinical Research Institute of Michigan, LLC - Troy, Troy, Michigan
  - Gastroenterology Associates of Western Michigan, Wyoming, Michigan
  - Kansas City Research Institute, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - St. Charles Clinical Research, Weldon Spring, Missouri
  - Montana Medical Research, Inc., Missoula, Montana
  - American Institute of Medical Research, Las Vegas, Nevada
  - Digestive Disease Specialists, Las Vegas, Nevada
  - Allied Health Clinical Research Organization, LLC (AHCRO) - Englewood, Englewood, New Jersey
  - Allied Health Clinical Research Organization, LLC (AHCRO) - Freehold, Freehold, New Jersey
  - Allied Health Clinical Research Organization, LLC (AHCRO) - Jackson, Jackson, New Jersey
  - NY Scientific, Brooklyn, New York
  - Smart Medical Research, Brooklyn, New York
  - Velocity Clinical Research - Syracuse, East Syracuse, New York
  - Tandem Clinical Research GI- New York, New York, New York
  - A1 Clinical Network, Richmond Hill, New York
  - OnSite Clinical Solutions, LLC, Charlotte, North Carolina
  - Atrium Health - Center for Digestive Health, Charlotte, North Carolina
  - Research Carolina Elite, LLC, Denver, North Carolina
  - Coastal Research Institute, LLC, Fayetteville, North Carolina
  - Cross Creek Medical, PA, Fayetteville, North Carolina
  - Triad Clinical Trials LLC, Greensboro, North Carolina
  - Peters Medical Research, High Point, North Carolina
  - Carolina's GI Research, Raleigh, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Remington Davis, Inc., Columbus, Ohio
  - DelRicht Clinical Research - Cincinnati, Mason, Ohio
  - Northshore Gastroenterology Research, LLC, Westlake, Ohio
  - Options Health Research, Tulsa, Oklahoma
  - Velocity Clinical Research, Medford, Oregon
  - Susquehanna Research Group, LLC, Harrisburg, Pennsylvania
  - Galen Medical Group - Downtown Gastroenterology Location, Chattanooga, Tennessee
  - WR ClinSearch, Chattanooga, Tennessee
  - DelRicht Clinical Research - Nashville, Henderson, Tennessee
  - North Hills Medical Research Inc. (North Hills Familiy Medicine), Arlington, Texas
  - Zenos Clinical Research, Dallas, Texas
  - Texas Gastro Research, LLC, El Paso, Texas
  - Houston Methodist Research Institute, Houston, Texas
  - Amir A Hassan, MD, PA, Houston, Texas
  - Care and Cure Clinic, Houston, Texas
  - Pioneer Research Solutions Inc., Houston, Texas
  - Epic Clinical Research, Lewisville, Texas
  - Texas Tech University Health Sciences Center, Lubbock, Texas
  - Biopharma Informatic, LLC, McAllen, Texas
  - DelRicht Clinical Research - McKinney, McKinney, Texas
  - Gastroenterology Research of San Antonio, San Antonio, Texas
  - A1 Clinical Network, Spring, Texas
  - HP Clinical Research (Val R. Hansen), Bountiful, Utah
  - Velocity Clinical Research - Salt Lake City, West Jordan, Utah
  - Manassas Clinical Research Center, Manassas, Virginia
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study website — https://www.gastroparesistrial.com/